Guy's, King's and St 25th Floor, Guy's Tower Thomas' Dental Institute Department London Bridge of Fixed and Removable Prosthodontics

Guy's Hospital London SE1 9RT Tel 0207 188 5390

Fax 0207 188 7486





## **Volunteer information sheet (Version 1) 1/12/13**

Title of project: Timing of dietary acid intake, brushing teeth and acid REC ref 14/WS/0015 NCT: NCT02449434 Investigator: Professor David Bartlett

Please complete this form after you have read the Information Sheet and/or listened to an explanation about the research

| Patient Identification: | Date |
|---|---|
| Thank you for considering taking part in this research. The person organising the research and/or a member of the clinical team who is trained for this purpose must explain the project before you agree to take part. | |
| If you have any questions arising from the Information Sheet or explanation given to you, please ask the researcher before you decide whether or not to join in. You will be given a copy of this Consent Form to keep and refer to at any time. | |
| I confirm that I have read and understand the information sheet dated (version 1) for the above study. | |
| | please initial each<br>box |
| I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being | |
| affected. I agree to take part in the above study. Name of Patient | |
| Name of Person taking consentSignature | |

 $\mbox{Guy's, King's and St} \qquad \mbox{$25^{th}$ Floor, Guy's Tower} \label{eq:Guy's}$ Thomas' Dental Institute Department London Bridge of Fixed and Removable Prosthodontics

Guy's Hospital London SE1 9RT Tel 0207 188 5390

Fax 0207 188 7486

